CLINICAL TRIAL: NCT02424968
Title: Post Transplant Infusion of Allogeneic CD8 Memory T-Cells as Consolidative Therapy After Non-myeloablative Allogeneic Hematopoietic Cell Transplantation in Patients With Leukemia and Lymphoma
Brief Title: CD8+ Memory T-Cells as Consolidative Therapy After Donor Non-myeloablative Hematopoietic Cell Transplant in Treating Patients With Leukemia or Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robert Lowsky (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Robert Lowsky, Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-33058; NCI-2015-00567 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 351 (IRB Number); BMT288 (Other: OnCore); P01CA049605 (NIH)
Record Dates: First submitted 2015-04-16; First posted 2015-04-23 (Estimated); Results first posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-05

CONDITIONS: Acute Myeloid Leukemia; B-Cell Non-Hodgkin Lymphoma; Chronic Lymphocytic Leukemia; Hodgkin Lymphoma; Myelodysplastic Syndrome; Myeloproliferative Neoplasm; T-Cell Non-Hodgkin Lymphoma
Keywords: Healthy Stem Cell Donor
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Hodgkin Disease; Myelodysplastic Syndromes; Myeloproliferative Disorders; Lymphoma, T-Cell | interventions — Antilymphocyte Serum; thymoglobulin; Cyclosporine; Cyclosporins; Mycophenolic Acid; Transplantation; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Infusion of Allogeneic CD8+ Memory T-cells (Experimental): All participants receive allogeneic CD8+ memory T-cells 30 to 60 days after standard non-myeloablative allogeneic hematopoietic cell transplant (aHCT).
  Interventions: Biological: Anti-Thymocyte Globulin; Drug: Cyclosporine; Drug: Mycophenolate Mofetil; Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplant; Biological: Allogeneic Cluster of Differentiation 8 (CD8)+ Memory T-cells; Radiation: Total Nodal Irradiation

INTERVENTIONS:
Biological: Anti-Thymocyte Globulin — Given per standard institutional practice
  Other Names: Antithymocyte Globulin; Antithymocyte Serum; ATG; ATGAM; ATS; Thymoglobulin
Drug: Cyclosporine — Given PO
  Other Names: 27-400; Ciclosporin; CsA; Cyclosporin; Cyclosporin A; Neoral; OL 27-400; Sandimmun; Sandimmune; SangCya
Drug: Mycophenolate Mofetil — Given PO
  Other Names: Cellcept; MMF
Procedure: Nonmyeloablative Allogeneic Hematopoietic Stem Cell Transplant — Undergo nonmyeloablative allogeneic HSCT
  Other Names: Non-myeloablative allogeneic transplant; Nonmyeloablative Stem Cell Transplant; NST; Peripheral Blood Stem Cell (PBSC) Transplant; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant
Biological: Allogeneic Cluster of Differentiation 8 (CD8)+ Memory T-cells — Receive CD8+ memory T-cells via IV
  Other Names: Allogeneic Lymphocytes; Tumor-Derived Lymphocyte
Radiation: Total Nodal Irradiation — Undergo TLI

SUMMARY:
This phase 2 trial studies how well cluster of differentiation 8 (CD8)+ memory T-cells work as a consolidative therapy following a donor non-myeloablative hematopoietic cell transplant in treating patients with leukemia or lymphoma. Giving total lymphoid irradiation and anti-thymocyte globulin before a donor hematopoietic cell transplant helps stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells (called graft-versus-host disease). Giving cyclosporine and mycophenolate mofetil after the transplant may stop this from happening. Once the donated stem cells begin working, the patient's immune system may see the remaining cancer cells as not belonging in the patient's body and destroy them. Giving an infusion of the donor's white blood cells, such as CD8+ memory T-cells, may boost this effect and may be an effective treatment to kill any cancer cells that may be left in the body (consolidative therapy).

DETAILED DESCRIPTION:
Participants undergo total lymphoid irradiation (TLI) on Days -11 to -7 and Days -4 to -1 and receive anti-thymocyte globulin (ATG) per standard institutional practice on Days -11 to -7. Patients also receive oral cyclosporine daily starting on Day -3, and will continue for at least 6 months post-transplant. Patients undergo standard non-myeloablative allogeneic HSCT on Day 0. Patients also receive oral mycophenolate mofetil daily beginning on Day 0 and continuing until Day 28. Participants receive an intravenous infusion of allogeneic cluster of differentiation 8 (CD8)+ memory T-cells over 10 to 20 minutes sometime between day 30 and day 60.

PRIMARY OBJECTIVES:

I. To determine the rate of conversion to full-donor chimerism (FDC) following a post-transplant infusion (Day 30-60) of freshly-enriched allogeneic CD8+ memory T-cells in patients with acute myeloid leukemia (AML), non-Hodgkin lymphoma (NHL), chronic lymphocytic leukemia (CLL), or Hodgkin lymphoma (HL), who received standard non-myeloablative total lymphoid irradiation (TLI) anti-thymocyte globulin (ATG) transplant conditioning.

SECONDARY OBJECTIVES:

I. To determine the risk of disease progression, overall and event free survival, and non-relapse mortality.

II. To determine the incidence of acute and chronic graft-versus-host disease (GVHD) following the infusion of allogeneic CD8+ memory T-cells.

OUTLINE:

Patients undergo TLI on days -11 to -7 and -4 to -1 and receive ATG per standard institutional practice on days -11 to -7. Patients also receive cyclosporine orally (PO) daily starting on day -3 and will continue for at least 6 months post-transplant. Patients undergo non-myeloablative allogeneic hematopoietic stem cell transplant (HSCT) on day 0. Patients also receive mycophenolate mofetil PO daily beginning on day 0 and continue until day 28. Based on the patient's status after the initial transplant, patients receive CD8+ memory T-cells intravenously (IV) over 10-20 minutes sometime between day 30 and day 60.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Must have a human leukocyte antigen (HLA)-matched or single allele-mismatched adult sibling serving as donor
* Must have a myeloid or lymphoid malignant disease that is treated with TLI and ATG reduced intensity conditioning for allogeneic transplant (any of the following AML, myelodysplastic syndrome [MDS], myeloproliferative disease [MPD], CLL, B or T-cell NHL, HL)
* Patients who due to age, pre-existing medical conditions, or, prior therapy are considered to be at high risk for regimen related toxicity associated with fully ablative transplant conditioning, and therefore reduced intensity conditioning is recommended
* Ability to understand and the willingness to sign a written informed consent document; patients must have signed informed consent to participate in the trial
* DONOR: Must be an HLA-matched or single allele mismatched sibling of enrolled transplant patient
* DONOR: Must be 18-75 years of age, inclusive
* DONOR: Must be in a state of general good health and have completed a donor evaluation with history, medical examination and standard blood tests within 35 days of starting the hematopoietic cell collection procedure; in order to fairly represent the interests of the donor, the donor evaluation and consent will be performed by a study team member other than the recipient's attending physician
* DONOR: Must have a white blood cell count > 3.5 x 10^9/liter, platelets > 150 x 10^9/liter and hematocrit > 35%
* DONOR: Must be capable of undergoing leukapheresis
* DONOR: Must be able to understand and sign informed consent
* DONOR: Must not be seropositive for HIV 1 and 2, hepatitis B surface antigen, hepatitis C antibody, human T-lymphotropic virus (HTLV) antibody, cytomegalovirus (CMV) immunoglobulin M (IgM), or rapid plasma reagin (RPR) (Treponema); donors with prior evidence of hepatitis B core antibody positivity will have a polymerase chain reaction (PCR) test done to evaluate for hepatitis B infection; donors with a positive hepatitis B PCR test are excluded
* DONOR: Females must not be pregnant or lactating
* DONOR: Must not have psychological traits or psychological or medical conditions which make them unlikely to tolerate the procedure
* DONOR: Must not have developed a new malignancy requiring chemotherapy or radiation in the interval since apheresis for initial hematocrit (HCT)
* PATIENT CRITERIA FOR PROCEEDING WITH CD8+ MEMORY T-CELL INFUSION:
* Patients must be beyond day 30 and before day 60 after transplant
* Patients must have evidence of mixed CD3 T-cell chimerism based on the day +28 (+/- 7 days) blood sample showing >= 5% and =< 95% donor type cells
* Patients must have no evidence of active graft-versus-host disease at the time of the CD8+ memory T-cell infusion; patients with a history of acute GVHD overall grade II based on skin only involvement or upper gastrointestinal (GI) tract involvement only will be eligible; patients with a history of liver or lower GI tract GVHD will not be eligible
* Patients must be on single immune suppression therapy with either tacrolimus or cyclosporine at the time of CD8+ memory T-cell infusion; prednisone at a physiologic dose of 5 mg per day or less is allowed
* Patients must have a Karnofsky performance status of >= 60% at the time of the CD8+ memory T-cell infusion
* Patients must not have an uncontrolled bacterial, fungal or viral infection, defined as progressive symptoms despite therapy, at the time of the CD8+ memory T-cell infusion; asymptomatic viremia is allowed
* Patients must have adequate organ function and performance status at the time of the CD8+ memory T-cell infusion, defined by the following:

  * Total bilirubin =< 4 mg/dL
  * SGOT or SGPT =< 4 x ULN
  * Creatinine =< 3 mg/dL or estimated creatinine clearance >= 40ml/min

Exclusion Criteria:

* Uncontrolled bacterial, viral or fungal infection defined as currently taking medication and progression of clinical symptoms
* Progressive hemato-lymphoid malignancy despite conventional therapy
* Acute leukemia not in remission
* Chronic myelogenous leukemia (CML)
* Active central nervous system (CNS) involvement of the underlying malignancy
* Human immunodeficiency virus (HIV) positive
* Pregnant or lactating
* Prior malignancy (EXCEPTION: diagnosed > 5 years ago without evidence of disease, OR treated =< 5 years ago but have a greater than 50% chance of life expectancy of >= 5 years for that malignancy)
* Have a psychiatric disorder(s) or psychosocial circumstance(s) which in the opinion of the primary physician would place the patient at an unacceptable risk from transplant
* Ejection fraction < 30%, or uncontrolled cardiac failure
* Diffusing capacity of the lung for carbon monoxide (DLCO) < 40% predicted
* Total bilirubin > 3 mg/dL
* Serum glutamic oxaloacetic transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) > 4 x upper limit of normal (ULN)
* Creatinine > 2 mg/dL and an estimated creatinine clearance =< 40 mL/min
* Poorly controlled hypertension despite multiple antihypertensive medication OR
* Karnofsky performance status (KPS) < 60%
* Note: Patients positive for hepatitis B and C will be evaluated on a case by case basis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-06; Primary Completion 2020-07-03 (Actual); Study Completion 2021-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Lowsky, Principal Investigator — Stanford University
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Infusion of Allogeneic CD8+ Memory T-cells
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Infusion of Allogeneic CD8+ Memory T-cells
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Full-dose Donor Chimerism (FDC)
Description: A measure of success for the therapeutic infusion of allogeneic transplantation of cluster of differentiation 8 (CD8+) memory T-cells is full-dose donor chimerism (FDC). This means to achieve ≥ 95% donor cells in either the CD3+ blood cell lineage or whole blood, within 90 days of the allogeneic CD8+ memory T-cell infusion. The outcome is reported as the number of participants that achieve FDC within 90 days, a number without dispersion.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Infusion of Allogeneic CD8+ Memory T-cells
Number analyzed (Participants) | 18
Participants | 12

2. Secondary Outcome: Event-free Survival (EFS
Description: Event-free survival (EFS) is defined as the number of transplant recipients of allogeneic cluster of differentiation 8 (CD8+) memory T-cells that remain alive at 12 months after transplant without disease relapse. Relapse is defined as bone marrow blasts > 5% . The outcome is expressed as the number of allogeneic CD8+ memory T-cell recipients remaining alive at 1 year after transplant without disease relapse, a number without dispersion.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Infusion of Allogeneic CD8+ Memory T-cells
Number analyzed (Participants) | 18
Participants | 15

3. Secondary Outcome: Incidence of Acute Graft vs Host Disease (GvHD)
Description: Occurrence of acute graft vs host disease (aGvHD) following the infusion of allogeneic transplantation of cluster of differentiation 8 (CD8+) memory T-cells will be assessed. The outcome is reported as the number of allogeneic CD8+ memory T-cell recipients who experience aGvHD within 30 days of the cellular infusion, a number without dispersion.
Time Frame: Up to 30 days post-infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Infusion of Allogeneic CD8+ Memory T-cells
Number analyzed (Participants) | 18
Participants | 1

4. Secondary Outcome: LOWSKY Grade 3 or Higher Toxicities
Description: Related adverse events, ie, toxicities, ≥ Grade 3 are significant considerations in the treatment of study participants receiving allogeneic transplantation of cluster of differentiation 8 (CD8+) memory T-cells. The outcome is reported as the number of allogeneic CD8+ memory T-cells transplant recipients who experienced ≥ Grade 3 toxicity within 60 days of infusion of the allogeneic transplantation of cluster of differentiation 8 (CD8+) memory T-cells, a number without dispersion.
Time Frame: Up to 60 days post-infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Infusion of Allogeneic CD8+ Memory T-cells
Number analyzed (Participants) | 18
Participants | 0

5. Secondary Outcome: Chronic Graft vs Host Disease (GvHD)
Description: The incidence of chronic graft vs host disease (cGvHD) following the infusion of allogeneic transplantation of cluster of differentiation 8 (CD8+) memory T-cells will be assessed. The outcome is reported as the number of allogeneic CD8+ memory T-cell recipients who experience cGvHD more 30 days but within 1 year of the cellular infusion, a number without dispersion.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Infusion of Allogeneic CD8+ Memory T-cells
Number analyzed (Participants) | 18
Participants | 2

6. Secondary Outcome: Non-relapse Mortality (NRM)
Description: Non-relapse mortality (NRM) is defined as death without known disease relapse or recurrence. The outcome is expressed as the number of allogeneic CD8+ memory T-cells tr. ansplant recipients whose cause of death was not disease relapse or recurrence, a number without dispersion
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Infusion of Allogeneic CD8+ Memory T-cells
Number analyzed (Participants) | 18
Participants | 1

7. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as remaining alive 12 months after the infusion of allogeneic cluster of differentiation 8 (CD8+) memory T-cells. The outcome is reported as the number of allogeneic CD8+ memory T-cell transplant recipients remaining alive at 12 months after the cellular infusion, a number without dispersion
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Infusion of Allogeneic CD8+ Memory T-cells
Number analyzed (Participants) | 18
Participants | 15

8. Secondary Outcome: Disease Progression (TDP)
Description: Whether or not the treated disease returns, known as disease progression or relapse, is a measure of treatment efficacy. Recipients of allogeneic transplantation of cluster of differentiation 8 (CD8+) memory T-cells were monitored for disease progression through 1 year after the cellular infusion. The outcome is reported as the number of allogeneic CD8+ memory T-cells recipients that experienced disease progression within 12 months (1 year).
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Infusion of Allogeneic CD8+ Memory T-cells
Number analyzed (Participants) | 18
Participants | 4

ADVERSE EVENTS:
Time Frame: 90 days
Description: Per protocol, Grade 1 to 2 adverse events were not collected. Grade 3 and higher adverse events were collected through 90 days (3 months) after the CD8+ memory T-cell infusion. Per protocol, policy, and practice, mortality (survival) is collected indefinitely.
Arm/Group | Infusion of Allogeneic CD8+ Memory T-cells
All-Cause Mortality (participants affected / at risk) | 3/18
Serious Adverse Events (participants affected / at risk) | 3/18
Other Adverse Events (participants affected / at risk) | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infusion of Allogeneic CD8+ Memory T-cells (N=18)
Lung Infection (Infections and infestations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-08-23): https://cdn.clinicaltrials.gov/large-docs/68/NCT02424968/Prot_SAP_001.pdf
  • Informed Consent Form (2020-03-11): https://cdn.clinicaltrials.gov/large-docs/68/NCT02424968/ICF_000.pdf